CLINICAL TRIAL: NCT01683357
Title: LONG-TERM RESULTS AFTER ONE-STAGE ULTRASOUND-GUIDED HEPATECTOMY IN PATIENTS WITH MULTIPLE BILOBAR COLORECTAL LIVER METASTASES: TOWARDS NEW CONCEPTS OF RADICAL RESECTION BY MEANS OF AN INTENTION TO TREAT ANALYSES
Brief Title: Prognosis of One-stage Hepatectomy for Bilobar Colorectal Metastases
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Director Liver Surgery Unit, Humanitas Cancer Center - Associate Professor, University of Milan, University of Milan
Other Study IDs: MTX-1STAGE LONG-TERM
Record Dates: First submitted 2012-09-04; First posted 2012-09-11 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Liver Metastases
Keywords: Liver Metastases; Surgery; Intraoperative Ultrasound
MeSH Terms: interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple Bilobar CLM: Patients selected for hepatectomy because carrier of multiple (> or = to 4), bilobar CLM
  Interventions: Procedure: Hepatectomy

INTERVENTIONS:
Procedure: Hepatectomy — Intraoperative ultrasound (IOUS) criteria for tumor-vessel relations let maximizing the preservation of the hepatic vascular skeleton. Contact between colorectal liver metastases and a major intrahepatic vessel is not by itself a criteria for vessel resection: tumor exposure is not contraindicated.
  If resection of a hepatic vein (HV), resection of the liver parenchyma drained by that vein is considered or not based on color-flow IOUS findings (hepatofugal blood flow in the feeding portal branch, evidence or not of communicating veins between adjacent HVs, evidence or not of accessory HVs).
  Parenchymal transection is performed under intermittent clamping by the Pringle maneuver. Drains are always inserted and a chest tube is inserted in patients undergoing thoracophrenolaparotomy.

SUMMARY:
It is not rare that two-stage hepatectomy for multiple bilobar colorectal liver metastases (CLM) be left incomplete because of disease progression or technical reasons. One-stage hepatectomy seems a feasible and safe alternative, however, long-term results are lacking. This study aims to provide evidence that one-stage hepatectomy compelling tumor exposure provides adequate long-term results with low risk of local recurrences.

DETAILED DESCRIPTION:
Eligibility Criteria The prospectively recruited cohort of patients herein analysed is the result of a policy for which those patients considered resectable and presenting 4 or more lesions, bilobar CLM were systematically approached in a one stage operation.

Patients were considered unresectable once there was concomitance of more than 3 lung metastases, diffuse peritoneal carcinomatosis, and/or extra-hilar lymph node metastasis.

Outcome measures The primary outcome was the feasibility on an intention-to-treat basis. To this purpose we studied the ratio between the number of patients surgically explored and those who effectively received resection.

The secondary outcome was the safety of the procedure. To this purpose we studied morbidity, mortality, amount of blood loss, rate of blood transfusions, and postoperative trend of liver function tests.

The tertiary outcome measure was the reliability of the procedure from an oncological standpoint. For this purpose we studied the following:

1. the rate of true local recurrence (cut-edge) after a minimum follow-up of 6 months;
2. the long-term follow-up, analysing the overall survival (survival after surgery), time to recurrence (survival without recurrence), and time to liver recurrence (survival without liver recurrence).
3. the overall survival compared with that based on an intention-to-treat criterion also including the outcome of those patients who met the inclusion criteria but resulted unresectable on exploration.

ELIGIBILITY:
Inclusion Criteria:

Those patients considered resectable and presenting 4 or more CLM, involving both liver lobes are systematically approached in a one stage operation.

Exclusion Criteria:

Patients carriers of more than 3 lung metastases, and/or diffuse peritoneal carcinomatosis, and/or extra-hilar lymph node metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with multiple (> or = to 4) and bilobar colorectal liver metastases
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2001-09; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
feasibility on an intention-to-treat basis | at the time of surgical intervention

SECONDARY OUTCOMES:
safety of the procedure | At 30 and 90 postoperative days
  Peroperative morbidity and mortality as classified according with Dindo-Clavien classification (see ref.); Amount of intraoperative blood loss and blood transfusions.

OTHER OUTCOMES:
reliability of the procedure from an oncological standpoint | 6-months of minimum follow-up for local recurrences; 5 years actuarial curves for overall survival and time to recurrence
  1. the rate of true local recurrence (cut-edge) after a minimum follow-up of 6 months;
  2. the long-term follow-up, analysing the overall survival (survival after surgery), time to recurrence (survival without recurrence), and time to liver recurrence (survival without liver recurrence).
  3. the overall survival compared with that based on an intention-to-treat criterion also including the outcome of those patients who met the inclusion criteria but resulted unresectable on exploration.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Torzilli, MD, PhD, Principal Investigator — University of Milan, Humanitas Cancer Center
Locations (1):
- Humanitas Cancer Center, Rozzano, Milano, Italy

REFERENCES:
- [Background] Wicherts DA, Miller R, de Haas RJ, Bitsakou G, Vibert E, Veilhan LA, Azoulay D, Bismuth H, Castaing D, Adam R. Long-term results of two-stage hepatectomy for irresectable colorectal cancer liver metastases. Ann Surg. 2008 Dec;248(6):994-1005. doi: 10.1097/SLA.0b013e3181907fd9. PMID 19092344
- [Background] Adam R, Laurent A, Azoulay D, Castaing D, Bismuth H. Two-stage hepatectomy: A planned strategy to treat irresectable liver tumors. Ann Surg. 2000 Dec;232(6):777-85. doi: 10.1097/00000658-200012000-00006. PMID 11088072
- [Background] Narita M, Oussoultzoglou E, Jaeck D, Fuchschuber P, Rosso E, Pessaux P, Marzano E, Bachellier P. Two-stage hepatectomy for multiple bilobar colorectal liver metastases. Br J Surg. 2011 Oct;98(10):1463-75. doi: 10.1002/bjs.7580. Epub 2011 Jun 28. PMID 21710481
- [Background] Jaeck D, Oussoultzoglou E, Rosso E, Greget M, Weber JC, Bachellier P. A two-stage hepatectomy procedure combined with portal vein embolization to achieve curative resection for initially unresectable multiple and bilobar colorectal liver metastases. Ann Surg. 2004 Dec;240(6):1037-49; discussion 1049-51. doi: 10.1097/01.sla.0000145965.86383.89. PMID 15570209
- [Background] Minagawa M, Makuuchi M, Torzilli G, Takayama T, Kawasaki S, Kosuge T, Yamamoto J, Imamura H. Extension of the frontiers of surgical indications in the treatment of liver metastases from colorectal cancer: long-term results. Ann Surg. 2000 Apr;231(4):487-99. doi: 10.1097/00000658-200004000-00006. PMID 10749608
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Result] Torzilli G, Procopio F, Botea F, Marconi M, Del Fabbro D, Donadon M, Palmisano A, Spinelli A, Montorsi M. One-stage ultrasonographically guided hepatectomy for multiple bilobar colorectal metastases: a feasible and effective alternative to the 2-stage approach. Surgery. 2009 Jul;146(1):60-71. doi: 10.1016/j.surg.2009.02.017. PMID 19541011
- [Result] Torzilli G, Montorsi M, Donadon M, Palmisano A, Del Fabbro D, Gambetti A, Olivari N, Makuuchi M. "Radical but conservative" is the main goal for ultrasonography-guided liver resection: prospective validation of this approach. J Am Coll Surg. 2005 Oct;201(4):517-28. doi: 10.1016/j.jamcollsurg.2005.04.026. PMID 16183489
- [Result] Torzilli G, Garancini M, Donadon M, Cimino M, Procopio F, Montorsi M. Intraoperative ultrasonographic detection of communicating veins between adjacent hepatic veins during hepatectomy for tumours at the hepatocaval confluence. Br J Surg. 2010 Dec;97(12):1867-73. doi: 10.1002/bjs.7230. Epub 2010 Aug 26. PMID 20799289
- [Result] Torzilli G, Montorsi M, Del Fabbro D, Palmisano A, Donadon M, Makuuchi M. Ultrasonographically guided surgical approach to liver tumours involving the hepatic veins close to the caval confluence. Br J Surg. 2006 Oct;93(10):1238-46. doi: 10.1002/bjs.5321. PMID 16953487
- [Result] Torzilli G, Palmisano A, Procopio F, Cimino M, Botea F, Donadon M, Del Fabbro D, Montorsi M. A new systematic small for size resection for liver tumors invading the middle hepatic vein at its caval confluence: mini-mesohepatectomy. Ann Surg. 2010 Jan;251(1):33-9. doi: 10.1097/SLA.0b013e3181b61db9. PMID 19858707
- [Result] Torzilli G, Procopio F, Donadon M, Del Fabbro D, Cimino M, Montorsi M. Safety of intermittent Pringle maneuver cumulative time exceeding 120 minutes in liver resection: a further step in favor of the "radical but conservative" policy. Ann Surg. 2012 Feb;255(2):270-80. doi: 10.1097/SLA.0b013e318232b375. PMID 21975322
- [Result] Torzilli G, Donadon M, Marconi M, Botea F, Palmisano A, Del Fabbro D, Procopio F, Montorsi M. Systematic extended right posterior sectionectomy: a safe and effective alternative to right hepatectomy. Ann Surg. 2008 Apr;247(4):603-11. doi: 10.1097/SLA.0b013e31816387d7. PMID 18362622
- [Result] Torzilli G, Del Fabbro D, Palmisano A, Donadon M, Bianchi P, Roncalli M, Balzarini L, Montorsi M. Contrast-enhanced intraoperative ultrasonography during hepatectomies for colorectal cancer liver metastases. J Gastrointest Surg. 2005 Nov;9(8):1148-53; discussion 1153-4. doi: 10.1016/j.gassur.2005.08.016. PMID 16269386